CLINICAL TRIAL: NCT06721754
Title: Diabetes Related Foot Ulcers with Negative Pressure Wound Therapy: a Randomized Controlled Trial
Brief Title: Diabetes Related Foot Ulcers with Negative Pressure Wound Therapy
Acronym: DIANE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Per-Henrik Randsborg, Professor MD, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 726929; 2024105 (Other Grant/Funding Number: South-Eastern Norway Regional Health Authority)
Record Dates: First submitted 2024-11-06; First posted 2024-12-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer; Negative Pressure Wound Treatment; Randomized Controlled Trial; Standard Wound Treatment; Amputation
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Wound Treatment (No Intervention)
- Negative Pressure Wound Treatment (Active Comparator)
  Interventions: Procedure: Negative Pressure Wound Treatment

INTERVENTIONS:
Procedure: Negative Pressure Wound Treatment — Negative Pressure Wound Treatment promotes healing by applying subatmospheric pressure to reduce inflammatory exudate and stimulate granulation tissue.
  Other Names: VAC
  Arms: Negative Pressure Wound Treatment

SUMMARY:
The goal of this study is to learn if the clinical effects of Negative Pressure Wound Therapy (NPWT) is better, worse or the same as standard wound care for patients with diabetic foot ulcers (DFUs).

The main questions it aims to answer are:

* Will there be a difference in the number of major amputations between the groups during the first year?
* Will one of the treatments require more surgeries and longer hospital stays?

All participants will:

* be treated with NPWT or standard wound care for their diabetic foot ulcer after surgery
* be followed closely at the out-patient clinic for one year after treatment

DETAILED DESCRIPTION:
Up to 34% of diabetic patients will develop a Diabetic Foot Ulcer (DFU) during their lifetime. Around one-third of patients with DFU end up with an amputation. The five-year mortality after major lower extremity amputation (LEA), defined as amputation at ankle level or above caused by a DFU, is 52% - 82%. The leading cause of the high mortality is an escalation of already established cardiovascular disease, kidney failure, and poor diabetes regulation. In addition, many amputees suffer from social isolation, depression, and lower quality of life. In 2021, 463 patients with diabetes were amputated in Norway. Approximately 33% of diabetes-related costs have been linked to the treatment of foot ulcers, the majority of which are related to inpatient hospital admissions. Data from England suggest that around 10% of hospital admissions among patients with diabetes were either for ulcer care or amputation. In the United States, $176 billion is spent annually on direct costs for diabetes care. One-third of this expenditure is lower-extremity-related, constituting a substantial cost to society.

A diabetic foot ulcer is challenging to treat and requires tedious care and often repeated surgical debridement, yet only two-thirds heal within 12 months. Both peripheral artery disease (PAD) and neuropathy are risk factors for the development of chronic foot ulceration in people with DM. Long healing times and one-year recurrence rates of over 20% have not improved in the past 20 years despite advances in wound care and revascularization techniques. The high prevalence of infection in DFU and the accompanying economic burden make it essential to develop cost-effective and limb-saving strategies to reduce the burden of DFU infection.

Negative Pressure Wound Therapy (NPWT)) also known as Vacuum Assisted Closure (VAC) therapy, was introduced two decades ago in an attempt to improve wound closure. NPWT aids wound healing by applying sub-atmospheric pressure to reduce inflammatory exudate and promote granulation tissue. It is widely used to manage complex wounds, including open fractures, burns, pressure ulcers, and diabetic foot ulcers. The application of NPWT therapy on chronic DFUs is recommended in several clinical guidelines, including the practical guidelines from the Wound Healing Society and the International Working Group on the Diabetic Foot. However, high-level documentation of the effect of NPWT therapy in the setting of DFU is lacking. Recently, several studies have examined the role of NPWT in the diabetic foot. The overall conclusion is that NPWT may have a positive effect, but the studies have methodological flaws and suffer a high risk of bias. It is, therefore, still being determined whether DFUs heal better with NPWT than with conventional wound care.

The investigators performed an internal quality audit of the treatment of DFU in our department. Despite following recommended procedures, including frequent use of NPWT, the investigators found that patients with DFU had extended hospital stays, underwent serial surgical revisions, and still required major LEA. In an attempt to reduce these complications, the investigators introduced a clinical pathway for patients with DFU to secure prioritized care, fast diagnosis, and treatment. Implementation of the clinical pathway reduced the number of major LEAs, number of surgical procedures, and length of hospital stays. Targeted and fast diagnosis, rapid initiation of treatment, and interdisciplinary collaboration with vascular surgery, infection medicine, and endocrinology were decisive for the outcome. In this new pathway, NPWT treatment was replaced with standard wound care. However, many different variables were altered at the same time. It is, therefore, unclear if the change from NPWT treatment to standard wound care influenced the outcome. Therefore, the purpose of this study is to compare the treatment of DFUs with either NPWT or standard wound care in terms of amputations and mortality, wound closure, hospital stay, and patient-reported outcomes. The study will clarify whether or not NPWT treatment helps treat chronic DFUs. The results will have a significant impact on a large patient group with high morbidity and mortality. The project will help define treatment recommendations that will reduce severe complications of DFU, such as LEA and wound recurrence, and improve the quality of life of diabetic patients. If successful, the project will reduce hospital stays and the number of surgical procedures, thus reducing healthcare costs for the institution and society. The project will obtain new knowledge on a frequently used intervention (NPWT), clarify its indications and limitations, and identify low-value care practices. The results will improve clinical practice and can be implemented in the healthcare system immediately. A prospective randomized controlled trial will be conducted at Akershus University Hospital. Patients referred to Akershus University Hospital will be invited and screened for eligibility. The surgeons will screen patients for trial eligibility by predetermined inclusion- and exclusion criteria and ensure that necessary examinations (MRI, CT, X-ray) have been done per protocol. Patients are invited to participate if all the inclusion criteria and none of the exclusion criteria are met. Eligible patients will receive an assessment by a dedicated healthcare worker, ensuring a thorough evaluation and sufficient reflection period for the patient. An independent third party will obtain informed consent to avoid undue pressure to participate in the study. Informed written and oral consent will be obtained. Patients will be recruited by all physicians who treat DFUs at the institution. A total of 50 patients will be included and randomized (25 patients in each trial arm).

NPWT-group: Patients allocated to NPWT will have the NPWT fitted at the end of wound debridement or partial amputation of the foot in the operating room. Negative pressure wound therapy is a closed, sealed system that applies negative pressure (suction) to the wound surface. Special foam padding is placed on or within the wound. A thin, clear, occlusive dressing seals the wound. A trackpad with suction connects to a canister to collect the fluid drainage. A special pump is used to apply negative pressure. Intermittent suction is maintained by connecting suction tubes from the wound dressing to a vacuum pump and liquid waste collector. The standard negative pressure is 125mmHg. Depending on clinical circumstances, the NPWT dressing is changed every 3-5 days, in theatre, bedside, or at the outpatient clinic, and discontinued as soon as possible. NPWT may be discontinued when the wound secretion is negligible and healthy granulation tissue is present.

Standard wound care group: After thorough debridement of the wound or partial amputation of the foot, dressings are applied to keep the base of the wound moist, control the exudation of the wound, avoid regular skin impregnation, and promote the formation of epithelium. Daily wound inspection and dressing changes are required when using moist compresses. The goal is secondary healing of the wound. After 2-4 days, if the wound is free of necrosis and pus, the dressing is changed to a hydrophobic-coated bacteria- and fungi binding wound dressing (Sorbact®) or an antibacterial silver dressing (Acticoat Ag 7) to cover the wound bed. The intact skin around the wound is covered by sterile cotton compresses or a self-adherent absorbent dressing (Mepore®). For both groups: Per-operatively, samples from pus, fluid, soft tissue, and bone (when osteomyelitis is suspected) are sent to microbiological culture. After sampling, intravenous antibiotics are initiated intravenously: Ekvacillin, Ciprofloxacin, Clindamycin, and Ciprofloxacin for patients with penicillin allergy. Treatment is adjusted according to microbiological growth and resistance patterns. The foot, ankle, and leg should be treated with compression stockings or elastic bandages for edemas. Patients may discontinue trial participation without having to provide any reason in accordance with the Helsinki Declaration. The data monitoring committee may discontinue follow-up in case of incorrect enrollment. Surgeons may also terminate a patient's trial participation if the patient develops other serious illnesses necessitating emergency surgery during the patient's follow-up period.

Withdrawal of trial participants: If the reason for withdrawal is voluntary discontinuation by the patient, no further data will be collected for that patient. However, data that has already been collected will be retained. All patients included will be accounted for in the trial flow diagram.

Patients who withdraw from the trial will be cared for and followed according to established clinical practice.

Criteria for LEA (primary outcome)

* Extensive plantar moist skin necrosis
* Excessive soft tissue necrosis
* In need of amputation of first and second metatarsal
* In need of amputation of >2 metatarsals
* Untreatable vascular occlusion and ischemia
* Untreatable osteomyelitis in the foot Adverse events
* Definition of Serious Adverse Events
* Death within 30 days postoperatively likely related to the DFU
* Major bleeding necessitating acute resuscitation, massive blood transfusion, or any additional vascular procedure to stop the bleeding.
* Any reoperation within 90 days of the index trial surgery due to deep wound infection, osteomyelitis, or sepsis
* Pulmonary embolism (PE)
* Acute myocardial infarction (AMI)
* Postoperative organ failure or worsening of pre-existing organ failure necessitating organ support or ICU stay.

Adverse events will be reported in electronic patient records according to clinical practice. During the hospital stay, an independent research coordinator will record complications and adverse effects consecutively.

Sample size calculation and statistical analysis: This study is focused on the primary outcome (amputation) at a one-year follow-up between the two treatment groups. For the power calculation, the investigators extrapolated the data from the introduction of the clinical pathway. When conducting the pilot, 11 % of LEAs (3 in 27 patients) were treated with standard wound care, compared to 65 % of LEAs (13 in 20 patients) treated with NPWT. For a conservative estimate, the investigators anticipated that there would be 55% LEA in the NPWT group compared to 15 % in the standard wound treatment group. The statistical power selected is 80%, and the accepted type I error rate is 5% (β =0.2, α = 0.05). Considering these assumptions and adding 20% for potential dropouts and mortality before one year, 25 (21+20%) patients are required in each group.

A statistician blinded to the group using delabeled data will analyze the primary and secondary outcomes. A study coordinator will register the adverse effects during the hospital stay and follow-up. Although a strictly conducted study regarding routines for completing the follow-up questionnaires, some loss to follow-up is expected. For missing data, imputation will be performed for the primary and secondary outcomes. Before the statistical analysis, the database will be locked for further data entry or alteration. A separate statistical analysis plan (SAP) will provide further details on imputation strategies and the planned statistical analyses. The SAP will be finalized, signed, and dated before the database lock and published at ClinicalTrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female above 18 years with a diabetic foot ulcer in need of surgical debridement or forefoot amputation

Exclusion Criteria:

* Previous leg amputation due to diabetes
* Unable to ambulate on feet
* Unlikely to adhere to treatment and/or follow-up
* Unable to complete questionnaire
* Active or ongoing cancer treatment
* In need of amputation at a higher level than metatarsal or more than two metatarsals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of lower extremity amputations | One year from inclusion
  The study will compare rates of lower extremity amputations within one year after two different treatments for diabetes related foot ulcers.

SECONDARY OUTCOMES:
Mortality | One year.
  Mortality rate during the study period.
Wound healing | One year.
  Wound healing during the study period.
Complications | One year.
  Rate of the following complications;
  * Death within 30 days postoperatively likely related to the DFU
  * Major bleeding necessitating acute resuscitation, massive blood transfusion, or any additional vascular procedure to stop the bleeding.
  * Any reoperation within 90 days of the index trial surgery, due to deep wound infection, osteomyelitis or sepsis
  * Pulmonary embolism (PE)
  * Acute myocardial infarction (AMI)
  * Postoperative organ failure or worsening of pre-existing organ failure necessitating organ support or ICU stay
Number of surgeries | One year.
  Number of surgeries during the study period.
Length of hospital stay | One year.
  Days of hospitalization during the study period.
Occupational status | At inclusion, 3, 6 and 12 months.
  Patient will report occupational status.
Patient-reported Outcome Measures (PROMS) | At inclusion, 3, 6 and 12 months.
  PROMS will be reported using:
  Health-related quality of life (EQ-5D-5L) The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  Foot and Ankle Ability Measure (FAAM) The FAAM is a patient-completed instrument that consists of an "Activities of Daily Living" subscale (21 scored items) and a "Sports" subscale (7 scored items) in which the response options are presented as 5-point Likert scales (range 4 to 0). Scores for each subscale range from 0% (least function) to 100% (most function).

CONTACTS AND LOCATIONS:
Overall Officials: Per-Henrik Randsborg, Professor; MD, Study Director — University Hospital, Akershus
Locations (1):
- Department of Orthopedic Surgery, Akershus University Hospital, Oslo, Nordbyhagen, Norway

IPD SHARING:
Plan to Share IPD: No
The data will be presented after collection and analysis in an article form.

REFERENCES:
- [Background] Schaper NC, van Netten JJ, Apelqvist J, Bus SA, Hinchliffe RJ, Lipsky BA; IWGDF Editorial Board. Practical Guidelines on the prevention and management of diabetic foot disease (IWGDF 2019 update). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3266. doi: 10.1002/dmrr.3266. PMID 32176447
- [Background] Schaper NC, van Netten JJ, Apelqvist J, Bus SA, Fitridge R, Game F, Monteiro-Soares M, Senneville E; IWGDF Editorial Board. Practical guidelines on the prevention and management of diabetes-related foot disease (IWGDF 2023 update). Diabetes Metab Res Rev. 2024 Mar;40(3):e3657. doi: 10.1002/dmrr.3657. Epub 2023 May 27. PMID 37243927
- [Background] Seidel D, Storck M, Lawall H, Wozniak G, Mauckner P, Hochlenert D, Wetzel-Roth W, Sondern K, Hahn M, Rothenaicher G, Kronert T, Zink K, Neugebauer E. Negative pressure wound therapy compared with standard moist wound care on diabetic foot ulcers in real-life clinical practice: results of the German DiaFu-RCT. BMJ Open. 2020 Mar 24;10(3):e026345. doi: 10.1136/bmjopen-2018-026345. PMID 32209619
- [Background] Armstrong DG, Lavery LA; Diabetic Foot Study Consortium. Negative pressure wound therapy after partial diabetic foot amputation: a multicentre, randomised controlled trial. Lancet. 2005 Nov 12;366(9498):1704-10. doi: 10.1016/S0140-6736(05)67695-7. PMID 16291063
- [Background] Woods TJ, Tesfay F, Speck P, Kaambwa B. Economic evaluations considering costs and outcomes of diabetic foot ulcer infections: A systematic review. PLoS One. 2020 Apr 30;15(4):e0232395. doi: 10.1371/journal.pone.0232395. eCollection 2020. PMID 32353082
- [Background] Kerr M, Rayman G, Jeffcoate WJ. Cost of diabetic foot disease to the National Health Service in England. Diabet Med. 2014 Dec;31(12):1498-504. doi: 10.1111/dme.12545. Epub 2014 Aug 1. PMID 24984759
- [Background] Hoffstad O, Mitra N, Walsh J, Margolis DJ. Diabetes, lower-extremity amputation, and death. Diabetes Care. 2015 Oct;38(10):1852-7. doi: 10.2337/dc15-0536. Epub 2015 Jul 22. PMID 26203063
- [Background] Armstrong DG, Swerdlow MA, Armstrong AA, Conte MS, Padula WV, Bus SA. Five year mortality and direct costs of care for people with diabetic foot complications are comparable to cancer. J Foot Ankle Res. 2020 Mar 24;13(1):16. doi: 10.1186/s13047-020-00383-2. PMID 32209136
- [Background] Thorud JC, Plemmons B, Buckley CJ, Shibuya N, Jupiter DC. Mortality After Nontraumatic Major Amputation Among Patients With Diabetes and Peripheral Vascular Disease: A Systematic Review. J Foot Ankle Surg. 2016 May-Jun;55(3):591-9. doi: 10.1053/j.jfas.2016.01.012. Epub 2016 Feb 19. PMID 26898398